CLINICAL TRIAL: NCT03101826
Title: Optimizing the Social Engagement System in Prader-Willi Syndrome: Insights From the Polyvagal Theory
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient resources
Sponsor: Indiana University (Other)
Collaborators: Latham Centers (Unknown)
Responsible Party: Principal Investigator, Stephen Porges, Distinguished University Scientist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1609337519
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Prader-Willi Syndrome
Keywords: Polyvagal Theory; Respiratory Sinus Arrhythmia; Heart rate; Social Behavior; Arginine Vasopressin; Dichotic Listening Tests; Oxytocin; Hyperacusis; Affect; Auditory perception; Sound spectrography
MeSH Terms: conditions — Prader-Willi Syndrome; Arrhythmia, Sinus; Social Behavior; Diabetes Insipidus; Hyperacusis

STUDY DESIGN:
Intervention Model Description: All participants will receive the active (filtered music) intervention.
Masking Description: No masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Filtered Music Intervention (Experimental): All participants will participate in pre-intervention assessments (6 months, 1 week prior) and post-intervention assessments (1 week, 1 month post). The Filtered Music Intervention (i.e., Listening Project Protocol) will last for 1 hour per day, for 5 consecutive days.
  Interventions: Behavioral: Listening Project Protocol

INTERVENTIONS:
Behavioral: Listening Project Protocol — The filtered music intervention will consist of listening to computer-altered acoustic stimulation, designed to modulate the frequency band of vocal music passed to the participant. The frequency characteristics of the acoustic stimulation are selected to emphasize the relative importance of specific frequencies in conveying the information embedded in human speech Modulation of the acoustic energy within the frequencies of human voice, similar to an exaggerated vocal prosody, are hypothesized to recruit and modulate the neural regulation of the middle ear muscles and to functionally reduce sound hypersensitivities and improve auditory processing.
  Other Names: Safe and Sound Protocol

SUMMARY:
The Polyvagal Theory focuses on how function and structure changed in the vertebrate autonomic nervous system during evolution. The theory is named for the vagus, a major cranial nerve that regulates bodily state. As a function of evolution, humans and other mammals have a "new" vagal pathway that links the regulation of bodily state to the control of the muscles of the face and head including the middle ear muscles. These pathways regulating body state, facial gesture, listening (i.e., middle ear muscles), and vocal communication collectively function as a Social Engagement System (SES). Because the Social Engagement System is an integrated system, interventions influencing one component of this system (e.g., middle ear muscles) may impact on the other components.

Individuals with Prader-Willi Syndrome (PWS) exhibit many behaviors that are consistent with a compromised Social Engagement System. Atypical function of the Social Engagement System results in problems associated with state regulation (e.g., impulsivity, tantrums, and difficulty with change in routine), ingestion (e.g., difficulties in sucking at birth, hyperphagia), coordination of suck/swallow/breathe, intonation of vocalizations, auditory processing and hypersensitivity, and socialization. We propose to confirm that several features of the behavioral phenotype of PWS may be explained within the context of a dysfunctional SES (Specific Aim I), which may be partially rehabilitated via an intervention designed as a 'neural exercise' of the SES (Specific Aim II).

Specific Aims:

Aim I: To demonstrate that children with PWS have atypical regulation of the SES. We hypothesize these effects will be manifested by dampened vagal regulation of the heart (low parasympathetic tone); poor middle ear muscle regulation resulting in auditory hypersensitivities and poor auditory processing; lack of voice intonation (prosody), and difficulties in accurately detecting the emotions of others.

Aim II: To demonstrate the effectiveness of the Listening Project Protocol (LPP) in decreasing the atypical features of the SES in adolescents with PWS. We hypothesize that individuals who complete the LPP will have improved vagal regulation of the heart, improved middle ear muscle regulation, increased voice intonation and improved ability to accurately detect the emotions of others.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be current residents at Latham Centers (LC) School in Brewster MA
2. Participants must meet criteria for Prader-Willi Syndrome
3. Participants must be between ages 13 - 25 years
4. Participants must have normal hearing
5. Participants must have normal vision (or corrected vision)

Exclusion Criteria:

1. Individuals with current (or a history of) heart disease
2. Individuals who are hearing-impaired
3. Individuals who are being treated for seizure disorder
4. Individuals who do not read/speak English
5. Individuals who are sight-impaired without correction

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Effect of Intervention on Autonomic regulation | Change from 1 week pre-intervention RSA to 1 month post-intervention
  Respiratory sinus arrhythmia (RSA)

SECONDARY OUTCOMES:
Effect of Intervention on Heart period | Change from 1 week pre-intervention heart period to 1 month post-intervention
  heart period
Effect of Intervention on Auditory processing | Change from 1 week pre-intervention Filtered Words to 1 month post-intervention
  Filtered Words subtest of SCAN
Effect of Intervention on Auditory processing | Change from 1 week pre-intervention Competing Words to 1 month post-intervention
  Competing Words subtest of SCAN
Effect of Intervention on Sensory Sensitivities | Change from 1 week pre-intervention BBC Sensory Scales to 1 month post-intervention
  BBC Sensory Scales (questionnaire)
Effect of Intervention on Latency to Affect recognition | Change from 1 week pre-intervention DARE (latency) to 1 month post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - latency
Effect of Intervention on Accuracy of Affect recognition | Change from 1 week pre-intervention DARE (accuracy) to 1 month post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - accuracy
Effect of Intervention on Prosody | Change from 1 week pre-intervention Prosody to 1 month post-intervention
  Analyses of vocal recordings
Effect of Intervention on Disruptive Behavior | Change from 1 week pre-intervention DBC to 1 month post-intervention
  Developmental Behavior Checklist (DBC) (questionnaire)
Effect of Intervention on Social behavior | Change from 1 week post-intervention LPP to 1 month post-intervention
  Listening Project Parent (LPP) Questionnaire
Effect of Intervention on Oxytocin | Change from 1 week pre-intervention oxytocin to 1 month post-intervention
  oxytocin levels derived from salivary sample
Effect of Intervention on Vasopressin | Change from 1 week pre-intervention vasopressin to 1 month post-intervention
  vasopressin levels derived from salivary sample

OTHER OUTCOMES:
Stability of Autonomic regulation | Change from 6 months pre-intervention RSA to 1 week pre-intervention
  Respiratory sinus arrhythmia (RSA)
Immediate effects of intervention on Autonomic regulation | Change from 1 week pre-intervention RSA to 1 week post-intervention
  Respiratory sinus arrhythmia (RSA)
Short-term effects of intervention on Autonomic regulation | Change from 1 week post-intervention RSA to 1 month post-intervention
  Respiratory sinus arrhythmia (RSA)
Stability of Heart period | Change from 6 months pre-intervention heart period to 1 week pre-intervention
  heart period
Immediate effects of intervention on Heart period | Change from 1 week pre-intervention heart period to 1 week post-intervention
  heart period
Short-term effects of intervention on Heart period | Change from 1 week post-intervention heart period to 1 month post-intervention
  heart period
Stability of Auditory processing | Change from 6 months pre-intervention Filtered Words to 1 week pre-intervention
  Filtered Words subtest of SCAN
Immediate effects of intervention on Auditory processing | Change from 1 week pre-intervention Filtered Words to 1 week post-intervention
  Filtered Words subtest of SCAN
Short-term effects of intervention on Auditory processing | Change from 1 week post-intervention Filtered Words to 1 month post-intervention
  Filtered Words subtest of SCAN
Stability of Auditory processing | Change from 6 months pre-intervention Competing Words to 1 week pre-intervention
  Competing Words subtest of SCAN
Immediate effects of intervention on Auditory processing | Change from 1 week pre-intervention Competing Words to 1 week post-intervention
  Competing Words subtest of SCAN
Short-term effects of intervention on Auditory processing | Change from 1 week post-intervention Competing Words to 1 month post-intervention
  Competing Words subtest of SCAN
Stability of Sensory Sensitivities | Change from 6 months pre-intervention BBC Sensory Scales to 1 week pre-intervention
  BBC Sensory Scales (questionnaire)
Stability of Latency to Affect recognition | Change from 6 months pre-intervention DARE latency to 1 week pre-intervention
  Dynamic Affect Recognition Evaluation (DARE) - latency
Immediate effects of intervention on Latency to Affect recognition | Change from 1 week pre-intervention DARE latency to 1 week post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - latency
Short-term effects of intervention on Latency to Affect recognition | Change from 1 week post-intervention DARE latency to 1 month post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - latency
Stability of Accuracy of Affect recognition | Change from 6 months pre-intervention DARE accuracy to 1 week pre-intervention
  Dynamic Affect Recognition Evaluation (DARE) - accuracy
Immediate effects of intervention on Accuracy of Affect recognition | Change from 1 week pre-intervention DARE accuracy to 1 week post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - accuracy
Short-term effects of intervention on Accuracy of Affect recognition | Change from 1 week post-intervention DARE accuracy to 1 month post-intervention
  Dynamic Affect Recognition Evaluation (DARE) - accuracy
Stability of Prosody | Change from 6 months pre-intervention prosody to 1 week pre-intervention
  Analyses of vocal recordings
Immediate effects of intervention on Prosody | Change from 1 week pre-intervention prosody to 1 week post-intervention
  Analyses of vocal recordings
Short-term effects of intervention on Prosody | Change from 1 week post-intervention prosody to 1 month post-intervention
  Analyses of vocal recordings
Stability of Disruptive behavior | Change from 6 months pre-intervention DBC to 1 week pre-intervention
  Developmental Behavior Checklist (DBC) (questionnaire)
Immediate effects of intervention on Disruptive behavior | Change from 1 week pre-intervention DBC to 1 week post-intervention
  Developmental Behavior Checklist (DBC) (questionnaire)
Short-term effects of intervention on Disruptive behavior | Change from 1 week post-intervention DBC to 1 month post-intervention
  Developmental Behavior Checklist (DBC) (questionnaire)
Stability of Oxytocin | Change from 6 months pre-intervention oxytocin to 1 week pre-intervention
  oxytocin levels derived from salivary sample
Stability of Vasopressin | Change from 6 months pre-intervention vasopressin to 1 week pre-intervention
  vasopressin levels derived from salivary sample

CONTACTS AND LOCATIONS:
Overall Officials: Stephen W Porges, PhD, Principal Investigator — Indiana University/Kinsey Institute
Locations (1):
- Latham Centers School, Brewster, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bal E, Harden E, Lamb D, Van Hecke AV, Denver JW, Porges SW. Emotion recognition in children with autism spectrum disorders: relations to eye gaze and autonomic state. J Autism Dev Disord. 2010 Mar;40(3):358-70. doi: 10.1007/s10803-009-0884-3. PMID 19885725
- [Background] Borg E, Counter SA. The middle-ear muscles. Sci Am. 1989 Aug;261(2):74-80. doi: 10.1038/scientificamerican0889-74. No abstract available. PMID 2667133
- [Background] Lewis GF, Furman SA, McCool MF, Porges SW. Statistical strategies to quantify respiratory sinus arrhythmia: are commonly used metrics equivalent? Biol Psychol. 2012 Feb;89(2):349-64. doi: 10.1016/j.biopsycho.2011.11.009. Epub 2011 Dec 3. PMID 22138367
- [Background] Porges SW. The polyvagal theory: phylogenetic substrates of a social nervous system. Int J Psychophysiol. 2001 Oct;42(2):123-46. doi: 10.1016/s0167-8760(01)00162-3. PMID 11587772
- [Background] Porges SW, Macellaio M, Stanfill SD, McCue K, Lewis GF, Harden ER, Handelman M, Denver J, Bazhenova OV, Heilman KJ. Respiratory sinus arrhythmia and auditory processing in autism: modifiable deficits of an integrated social engagement system? Int J Psychophysiol. 2013 Jun;88(3):261-70. doi: 10.1016/j.ijpsycho.2012.11.009. Epub 2012 Nov 29. PMID 23201146
- [Background] Porges SW, Bazhenova OV, Bal E, Carlson N, Sorokin Y, Heilman KJ, Cook EH, Lewis GF. Reducing auditory hypersensitivities in autistic spectrum disorder: preliminary findings evaluating the listening project protocol. Front Pediatr. 2014 Aug 1;2:80. doi: 10.3389/fped.2014.00080. eCollection 2014. PMID 25136545